CLINICAL TRIAL: NCT01218776
Title: International Survey of Acute Coronary Syndromes
Acronym: ISACS
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Raffaele Bugiardini, Principal Investigator, University of Bologna
Other Study IDs: ISACS-TC 1
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome; Unstable Angina Pectoris; Myocardial Infarction; Coronary Disease
Keywords: Acute Coronary Syndrome, Eastern Europe, Therapies
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Myocardial Infarction; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells,
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male, Female, Kidney Disease, Elderly: Non-interventional patient registry

SUMMARY:
The International Registry of Acute Coronary Syndromes registry study (ISACS) is both a retrospective and prospective study which was designed in order to obtain data of patients with acute coronary syndromes, and herewith control and optimize internationally guideline-recommended therapies in these countries

DETAILED DESCRIPTION:
Aims of this survey study are (1) documentation of the characteristics of all patients presenting to the ISACS centers with STEMI or NSTEMI (2) documentation of in-hospital outcome, and outcome rates at 6 month and 1 year, (3) documentation of invasive procedures and procedure-associated complications (4) documentation of therapeutic regimens and investigation conformity of treatment with already established guidelines.

Investigators:

ISACS Administrative Committee:

Raffaele Bugiardini (Italy-Principal Investigator) Lina Badimon (Spain) Olivia Manfrini (Italy- Project Coordinator) Edina Cenko (Italy-Center Coordinator)

Steering Committee:

Mirza Dilic (Bosnia and Herzegovina), Asen Goudev (Bulgaria), Davor Milicic (Croatia), Raffaele Bugiardini, Edina Cenko and Olivia Manfrini (Italy) Gani Bajraktari (Kosovo), Andrejs Erglis and Ilja Zakke (Latvia), Remigius Zaliunas and Olivija Gustiene (Lithuania), Sasko Kedev and Marija Vavlukis (North Macedonia), Mihail Popovici (Moldova), Maria Dorobantu (Romania), Zorana Vasiljevic (Serbia), Eva Goncalvesova and Martin Studenkan (Slovakia) , Alexander N. Parkhomenko (Ukraine) , Christopher P Gale (United Kingdom).

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndromes

Exclusion Criteria:

* under age or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted with a diagnosis of acute coronary syndromes.
Sampling Method: Probability Sample
Enrollment: 36000 (Estimated)
Dates: Start 2010-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All causes mortality | 30 days, 6 months, 1 year
  All causes mortality

SECONDARY OUTCOMES:
Cardiovascular mortality | 30 days, 6 months, 1 year
  Cardiovascular mortality
Recurrent myocardial infarction | 30 days, 6 months, 1year
  Recurrent myocardial infarction
Pharmacogenetic and cardiovascular genetic studies associated to clinical outcomes | 6 month, 1 year
  Pharmacogenetic and cardiovascular genetic studies associated to clinical outcomes
Adherence to internationally guideline recommended therapies across the participating countries | discharge, 6 months, 1 year
  Adherence to internationally guideline recommended therapies across the participating

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Bugiardini, MD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Bugiardini R, Badimon L , Manfrini O. Rationale and design of the ISACS-TC (International Survey of Acute Coronary Syndromes in Transitional Countries) project. Eur Heart J Suppl. 2014;16 (suppl A): A1-A6 DOI: http://dx.doi.org/10.1093/eurheartj/sut002. First published online: 10 January 2014
- [Result] Bugiardini R, Dorobantu M, Vasiljevic Z, Kedev S, Knezevic B, Milicic D, Calmac L, Trninic D, Daullxhiu I, Cenko E, Ricci B, Puddu PE, Manfrini O, Koller A, Badimon L; ISACS-TC Investigators. Unfractionated heparin-clopidogrel combination in ST-elevation myocardial infarction not receiving reperfusion therapy. Atherosclerosis. 2015 Jul;241(1):151-6. doi: 10.1016/j.atherosclerosis.2015.04.794. Epub 2015 Apr 27. PMID 25988359
- [Result] Bugiardini R, Cenko E, Ricci B, Vasiljevic Z, Dorobantu M, Kedev S, Vavlukis M, Kalpak O, Puddu PE, Gustiene O, Trninic D, Knezevic B, Milicic D, Gale CP, Manfrini O, Koller A, Badimon L. Comparison of Early Versus Delayed Oral beta Blockers in Acute Coronary Syndromes and Effect on Outcomes. Am J Cardiol. 2016 Mar 1;117(5):760-7. doi: 10.1016/j.amjcard.2015.11.059. Epub 2015 Dec 13. PMID 26778165
- [Result] Manfrini O, Dorobantu M, Vasiljevic Z, Kedev S, Knežević B, Miličić D, Dilic M, Trninic D, Daullxhiu I, Gustienė O, Ricci B, Martelli I, Cenko E, Koller A, Badimon L, Bugiardini R. Acute coronary syndrome in octogenarian patients: results from the international registry of acute coronary syndromes in transitional countries (ISACS-TC) registry. Eur Heart J Suppl.2014;16 (suppl A): A87-A94. DOI: http://dx.doi.org/10.1093/eurheartj/sut019. First published online: 10 January 2014
- [Result] Cenko E, Ricci B, Kedev S, Vasiljevic Z, Dorobantu M, Gustiene O, Knezevic B, Milicic D, Dilic M, Trninic D, Smith F, Manfrini O, Badimon L, Bugiardini R. Reperfusion therapy for ST-elevation acute myocardial infarction in Eastern Europe: the ISACS-TC registry. Eur Heart J Qual Care Clin Outcomes. 2016 Jan 1;2(1):45-51. doi: 10.1093/ehjqcco/qcv025. PMID 29474588
- [Result] Dorobantu M, Tautu O.-F, Fruntelata A, Calmac L, Tatu-Chitoiu G, Bataila V, Dimulescu D, Craiu E, Nanea T, Istvan A, Babes K, Macarie C, Militaru C, Cenko E, Manfrini O. Hypertension and acute coronary syndromes in Romania: Data from the ISACS-TC registry. Eur Heart J Suppl (2014) 16 (suppl A): A20-A27 DOI: http://dx.doi.org/10.1093/eurheartj/sut006 First published online: 10 January 2014
- [Result] Vasiljevic Z, Krljanac G, Davidovic G, Panic G, Radovanovic S, Mickovski N, Srbljak N, Markovic-Nikolic N, Curic-Petkovic S, Panic M, Cenko E, Manfrini O, Martelli I, Koller A, Badimon L, Bugiardini R. Gender differences in case fatality rates of acute myocardial infarction in Serbia. Eur Heart J Suppl (2014) 16 (suppl A): A48-A55 DOI: http://dx.doi.org/10.1093/eurheartj/sut012 First published online: 10 January 2014
- [Result] Trninic D, Dilic M, Vasiljevic Z, Kulic M, Srdić S, Dobrijević N, Sabanovic-Bajramovic N, Begic A, Kukavica N, Vukcevic V, Davidovic G, Panic G, Saric J, Zrnic M, Matic I, Trifunovic N, Martelli I, Cenko E, Manfrini O, Koller A, Badimon L, Bugiardini R. Clinical profile of patients with no-reperfusion therapy in Bosnia and Herzegovina and Serbia. Eur Heart J Suppl (2014) 16 (suppl A): A67-A73 DOI: http://dx.doi.org/10.1093/eurheartj/sut015 First published online: 10 January 2014
- [Result] Manfrini O, Ricci B, Cenko E, Dorobantu M, Kalpak O, Kedev S, Knezevic B, Koller A, Milicic D, Vasiljevic Z, Badimon L, Bugiardini R; ISACS-TC Investigators. Association between comorbidities and absence of chest pain in acute coronary syndrome with in-hospital outcome. Int J Cardiol. 2016 Aug;217 Suppl:S37-43. doi: 10.1016/j.ijcard.2016.06.221. Epub 2016 Jun 28. PMID 27381858
- [Result] Calmac L, Bataila V, Ricci B, Vasiljevic Z, Kedev S, Gustiene O, Trininic D, Knezevic B, Milicic D, Dilic M, Manfrini O, Cenko E, Badimon L, Bugiardini R, Scafa-Udriste A, Tautu O, Dorobantu M. Factors associated with use of percutaneous coronary intervention among elderly patients presenting with ST segment elevation acute myocardial infarction (STEMI): Results from the ISACS-TC registry. Int J Cardiol. 2016 Aug;217 Suppl:S21-6. doi: 10.1016/j.ijcard.2016.06.227. Epub 2016 Jun 29. PMID 27381859
- [Result] Bugiardini R, Badimon L; ISACS-TC Investigators and Coordinators. The International Survey of Acute Coronary Syndromes in Transitional Countries (ISACS-TC): 2010-2015. Int J Cardiol. 2016 Aug;217 Suppl:S1-6. doi: 10.1016/j.ijcard.2016.06.219. Epub 2016 Jun 28. PMID 27386758
- [Result] Cenko E, Ricci B, Kedev S, Kalpak O, Calmac L, Vasiljevic Z, Knezevic B, Dilic M, Milicic D, Manfrini O, Koller A, Dorobantu M, Badimon L, Bugiardini R. The no-reflow phenomenon in the young and in the elderly. Int J Cardiol. 2016 Nov 1;222:1122-1128. doi: 10.1016/j.ijcard.2016.07.209. Epub 2016 Aug 2. PMID 27499222
- [Result] Ricci B, Manfrini O, Cenko E, Vasiljevic Z, Dorobantu M, Kedev S, Davidovic G, Zdravkovic M, Gustiene O, Knezevic B, Milicic D, Badimon L, Bugiardini R. Primary percutaneous coronary intervention in octogenarians. Int J Cardiol. 2016 Nov 1;222:1129-1135. doi: 10.1016/j.ijcard.2016.07.204. Epub 2016 Aug 2. PMID 27506888
- [Result] Cenko E, Ricci B, Kedev S, Vasiljevic Z, Dorobantu M, Gustiene O, Knezevic B, Milicic D, Dilic M, Manfrini O, Koller A, Badimon L, Bugiardini R. Invasive versus conservative strategy in acute coronary syndromes: The paradox in women's outcomes. Int J Cardiol. 2016 Nov 1;222:1110-1115. doi: 10.1016/j.ijcard.2016.07.211. Epub 2016 Jul 30. PMID 27514628
- [Result] Bugiardini R, Ricci B, Cenko E, Vasiljevic Z, Kedev S, Davidovic G, Zdravkovic M, Milicic D, Dilic M, Manfrini O, Koller A, Badimon L. Delayed Care and Mortality Among Women and Men With Myocardial Infarction. J Am Heart Assoc. 2017 Aug 21;6(8):e005968. doi: 10.1161/JAHA.117.005968. PMID 28862963
- [Result] Ricci B, Cenko E, Vasiljevic Z, Stankovic G, Kedev S, Kalpak O, Vavlukis M, Zdravkovic M, Hinic S, Milicic D, Manfrini O, Badimon L, Bugiardini R. Acute Coronary Syndrome: The Risk to Young Women. J Am Heart Assoc. 2017 Dec 22;6(12):e007519. doi: 10.1161/JAHA.117.007519. PMID 29273636
- [Result] Cenko E, Yoon J, Kedev S, Stankovic G, Vasiljevic Z, Krljanac G, Kalpak O, Ricci B, Milicic D, Manfrini O, van der Schaar M, Badimon L, Bugiardini R. Sex Differences in Outcomes After STEMI: Effect Modification by Treatment Strategy and Age. JAMA Intern Med. 2018 May 1;178(5):632-639. doi: 10.1001/jamainternmed.2018.0514. PMID 29630703
- [Result] Cenko E, van der Schaar M, Yoon J, Kedev S, Valvukis M, Vasiljevic Z, Asanin M, Milicic D, Manfrini O, Badimon L, Bugiardini R. Sex-Specific Treatment Effects After Primary Percutaneous Intervention: A Study on Coronary Blood Flow and Delay to Hospital Presentation. J Am Heart Assoc. 2019 Feb 19;8(4):e011190. doi: 10.1161/JAHA.118.011190. PMID 30764687
- [Result] Cenko E, van der Schaar M, Yoon J, Manfrini O, Vasiljevic Z, Vavlukis M, Kedev S, Milicic D, Badimon L, Bugiardini R. Sex-Related Differences in Heart Failure After ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2019 Nov 12;74(19):2379-2389. doi: 10.1016/j.jacc.2019.08.1047. PMID 31699278
- [Result] Bugiardini R, Yoon J, Kedev S, Stankovic G, Vasiljevic Z, Milicic D, Manfrini O, van der Schaar M, Gale CP, Badimon L, Cenko E. Prior Beta-Blocker Therapy for Hypertension and Sex-Based Differences in Heart Failure Among Patients With Incident Coronary Heart Disease. Hypertension. 2020 Sep;76(3):819-826. doi: 10.1161/HYPERTENSIONAHA.120.15323. Epub 2020 Jul 13. PMID 32654558
- [Result] Bugiardini R, Yoon J, Mendieta G, Kedev S, Zdravkovic M, Vasiljevic Z, Milicic D, Manfrini O, van der Schaar M, Gale CP, Bergami M, Badimon L, Cenko E. Reduced Heart Failure and Mortality in Patients Receiving Statin Therapy Before Initial Acute Coronary Syndrome. J Am Coll Cardiol. 2022 May 24;79(20):2021-2033. doi: 10.1016/j.jacc.2022.03.354. PMID 35589164
- [Result] Bergami M, Cenko E, Yoon J, Mendieta G, Kedev S, Zdravkovic M, Vasiljevic Z, Milicic D, Manfrini O, van der Schaar M, Gale CP, Badimon L, Bugiardini R. Statins for primary prevention among elderly men and women. Cardiovasc Res. 2022 Nov 10;118(14):3000-3009. doi: 10.1093/cvr/cvab348. PMID 34864917
- [Result] Bugiardini R, Cenko E, Yoon J, van der Schaar M, Kedev S, Gale CP, Vasiljevic Z, Bergami M, Milicic D, Zdravkovic M, Krljanac G, Badimon L, Manfrini O. Concerns about the use of digoxin in acute coronary syndromes. Eur Heart J Cardiovasc Pharmacother. 2022 Aug 11;8(5):474-482. doi: 10.1093/ehjcvp/pvab055. PMID 34251454
- [Result] Bugiardini R, Pavasovic S, Yoon J, van der Schaar M, Kedev S, Vavlukis M, Vasiljevic Z, Bergami M, Milicic D, Manfrini O, Cenko E, Badimon L. Aspirin for primary prevention of ST segment elevation myocardial infarction in persons with diabetes and multiple risk factors. EClinicalMedicine. 2020 Sep 20;27:100548. doi: 10.1016/j.eclinm.2020.100548. eCollection 2020 Oct. PMID 33150322
- [Result] Manfrini O, Yoon J, van der Schaar M, Kedev S, Vavlukis M, Stankovic G, Scarpone M, Milicic D, Vasiljevic Z, Badimon L, Cenko E, Bugiardini R. Sex Differences in Modifiable Risk Factors and Severity of Coronary Artery Disease. J Am Heart Assoc. 2020 Oct 20;9(19):e017235. doi: 10.1161/JAHA.120.017235. Epub 2020 Sep 28. PMID 32981423
- [Derived] Cenko E, Bergami M, Yoon J, Vadala G, Kedev S, Kostov J, Vavlukis M, Vraynko E, Milicic D, Vasiljevic Z, Zdravkovic M, Galassi AR, Manfrini O, Bugiardini R. Age and sex differences in the efficacy of early invasive strategy for non-ST-elevation acute coronary syndrome: A comparative analysis in stable patients. Am J Prev Cardiol. 2025 Mar 29;22:100984. doi: 10.1016/j.ajpc.2025.100984. eCollection 2025 Jun. PMID 40256411
- [Derived] Fabin N, Cenko E, Bergami M, Yoon J, Vadala G, Mendieta G, Kedev S, Kostov J, Vavlukis M, Vraynko E, Milicic D, Vasiljevic Z, Zdravkovic M, Badimon L, Galassi AR, Manfrini O, Bugiardini R. Early coronary revascularization among 'stable' patients with non-ST-segment elevation acute coronary syndromes: the role of diabetes and age. Cardiovasc Res. 2024 Dec 14;120(16):2064-2077. doi: 10.1093/cvr/cvae190. PMID 39196713
- [Derived] Vasiljevic-Pokrajcic Z, Mickovski N, Davidovic G, Asanin M, Stefanovic B, Krljanac G, Radosavljevic-Radovanovic M, Radovanovic N, Lasica R, Milanovic S, Bjekic J, Majstorovic-Stakic M, Trifunovic D, Karadzic A, Rajic D, Milosevic A, Zdravkovic M, Saric J, Bugiardini R. Sex and age differences and outcomes in acute coronary syndromes. Int J Cardiol. 2016 Aug;217 Suppl:S27-31. doi: 10.1016/j.ijcard.2016.06.217. Epub 2016 Jun 27. PMID 27395070